CLINICAL TRIAL: NCT06235437
Title: A Phase 1, First-in-Human, Open-label, Doseescalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ASD141 in Subjects With Advanced Solid Tumors
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ASD141
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascendo Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABU001
Record Dates: First submitted 2024-01-18; First posted 2024-02-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Subjects will receive one of 8 dose levels of ASD141 (0.01, 0.03, 0.1, 0.3, 1, 3, 10, and 30 mg/kg) once every week (QW) in a 28-day cycle. BOIN design with accelerated titration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASD141 (Experimental): IV, Monotherapy
  Interventions: Biological: ASD141

INTERVENTIONS:
Biological: ASD141 — Subjects will receive one of 8 dose levels of ASD141.

SUMMARY:
This is a Phase I study designed to evaluate if ASD141 is safe, tolerable, and efficacious in participants with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, first-in-human (FIH), open-label, non-randomized, dose escalation study of ASD141 to evaluate safety, tolerability, and preliminary anti-tumor activity of ASD141 in subjects with advanced solid tumors. The study includes 8 dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily agreed to participate by giving written informed consent.
* Male or female ≥ 18 years of age on the day of signing informed consent.
* Has a histologically or cytologically confirmed metastatic solid tumor for which there is no available therapy that is expected to convey clinical benefit.
* Has at least one measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Subjects must have a performance status of ≤ 1 on the ECOG performance scale.
* Subjects must have adequate organ function as indicated by the following laboratory values. Hematological Neutrophil Count (ANC) ≥ 1,500 /µL (mm3) Platelets ≥ 100,000 /µL (mm3) Hemoglobin ≥ 9 g/dL Renal estimated GFR (non-indexed)* ≥ 50 mL/min Hepatic Serum total bilirubin ≤ 1.5X ULN OR Direct bilirubin ≤ 1.5X ULN for subjects with total bilirubin levels > 1.5 ULN; ≤ 3X ULN for subjects with hepatoma or Gilbert's disease AST and ALT ≤ 2.5X ULN OR ≤ 5X ULN for subjects with active liver metastases and primary hepatoma Coagulation International normalized ratio (INR) ≤ 1.5X ULN Activated partial thromboplastin time (aPTT) ≤ 1.5X ULN
* QTcF < 480 msec
* Female subject of childbearing potential has a negative serum pregnancy test.
* Female subjects of childbearing potential and male subjects must be willing to use adequate contraceptive methods during the study treatment and for at least 90 days after the last dose of study treatment. Acceptable contraceptive methods include implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, diaphragm with spermicide, cervical cap with spermicide, male or female condom with spermicide or a partner who is sterile. Spermicides alone are not an acceptable method of contraception.
* Has provided a tumor tissue sample (latest archival or newly obtained core or excisional biopsy of a tumor lesion).

Exclusion Criteria:

* Has had curative radiotherapy, investigational or approved cancer therapy (e.g., chemotherapy, biologics, hormone [e.g., tamoxifen, leuprolide]) within 2 weeks or 5 halflives (whichever is shorter) prior to the first dose of study treatment.
* Has not recovered to Common Toxicity Criteria for Adverse Events (CTCAE) Grade 1 or better from the adverse events due to previous anti-cancer therapy prior to the first dose of study treatment, with the exception of alopecia and ≤ Grade 2 peripheral neuropathy.
* Has used an investigational device or has had major surgery within 4 weeks prior to the first dose of study treatment.
* Has received previous treatment with another agent targeting the CD11b receptor.
* Is expected to require any other forms of antineoplastic therapy while participating in the study.
* Is on chronic systemic steroid therapy in excess of replacement doses or on any other form of immunosuppressive medication.
* Has a history of a previous additional malignancy unless potentially curative treatment has been completed with no evidence of malignancy for at least 2 years prior to the first dose of study treatment. Subjects with carcinoma in situ of any origin are eligible.
* Has active central nervous system (CNS) metastases and/or carcinomatous meningitis.

Subjects with CNS metastases are eligible if they are asymptomatic (including those who have never received any treatment) and not requiring concurrent treatment, including but not limited to surgery, radiation, corticosteroids and/or anticonvulsants to treat CNS metastases.

* Has an active autoimmune disease.
* Has an acute active infection requiring systemic treatment.
* Has interstitial lung disease.
* Has active or a history of non-infectious pneumonitis requiring steroids.
* Has symptomatic ascites or pleural effusion.
* Has previously had a hematopoietic stem cell transplant or solid organ transplant.
* Is known to have active chronic or acute Hepatitis B; however, subjects with HBV DNA

  ≤ 2000 IU/mL with or without antiviral therapy are eligible.
* Has received a live-virus vaccine within 4 weeks prior to the first dose of study treatment.
* Has received an mRNA vaccine within 4 months prior to the first dose of study treatment.
* Has any of the following condition within 3 months of the first dose of study treatment:

deep vein thrombosis, pulmonary embolism, myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack.

* Has a history of allergic reactions to any of the components of ASD141 Injection (i.e., sodium citrate, sucrose, and polysorbate 80).
* Has a history of severe hypersensitivity or anaphylactic reactions (e.g., shock, asthma etc.).
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicity | 28 days
  Frequency of dose-limiting toxicity (DLT) at each dose level
Percentage of participants with adverse events (AEs) and serious AEs (SAEs), vital signs, and abnormal laboratory parameters | Dose Escalation (From the time of informed consent until 90 days after the last dose of ASD141)
  Frequency, type, severity, and relationship to ASD141 of adverse events (AEs)

SECONDARY OUTCOMES:
Plasma Cmax | Dose Escalation (From the time of informed consent until 90 days after the last dose of ASD141)
  maximum measured concentration of ASD141 in plasma
Plasma AUClast | Dose Escalation (From the time of informed consent until 90 days after the last dose of ASD141)
  area under the plasma concentration-time curve of ASD141 from hour 0 to last sample with measurable plasma concentrations
Plasma AUCinfinity | Dose Escalation (From the time of informed consent until 90 days after the last dose of ASD141)
  area under the plasma concentration-time curve of ASD141 in plasma over the time interval from 0 extrapolated to infinity
Plasma t1/2 | Dose Escalation (From the time of informed consent until 90 days after the last dose of ASD141)
  terminal half-life of ASD141 in plasma
Plasma tmax | Dose Escalation (From the time of informed consent until 90 days after the last dose of ASD141)
  Time of the maximum observed ASD141 concentration
anti-drug antibodies (ADAs) | Dose Escalation (From the time of informed consent until 90 days after the last dose of ASD141)
  Presence or absence of anti-drug antibodies (ADAs) against ASD141
Objective response rate | Dose Escalation (From first dose of ASD141 to progressive disease (PD) or death in the absence of disease progression (approximately 1 year)
  Percentage of participants with a confirmed CR or PR according to RECIST v1.1
Progressive free survival | Dose Escalation (From first dose of ASD141 to progressive disease (PD) or death in the absence of disease progression (approximately 1 year)
  The time from first dose of study intervention until the date of objective disease progression or death in the absence of disease progression
Disease control rate | Dose Escalation (From first dose of ASD141 to progressive disease (PD) or death in the absence of disease progression (approximately 1 year)
  Percentage of participants who have a best objective response of confirmed CR or PR or who have SD lasting for at least a certain time of period after start of treatment
Duration of response | Dose Escalation (From first dose of ASD141 to progressive disease (PD) or death in the absence of disease progression (approximately 2 year)
  The time from first response according to RECIST v1.1 and iRECIST v1.1 until progression or death in the absence of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Min Yeh, M.D. PhD., Principal Investigator — National Cheng-Kung University Hospital
Locations (2):
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No